CLINICAL TRIAL: NCT00126646
Title: Phase I Study of BL22, A Recombinant Immunotoxin for Chronic Lymphocytic Leukemia and CD22+ Lymphomas
Brief Title: BL22 Immunotoxin in Treating Patients With Refractory Chronic Lymphocytic Leukemia, Prolymphocytic Leukemia, or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Robert Kreitman , MD, NCI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000438672; NCI-05-C-0171; NCI-P6620; NCI-5336; NCT00114751 (obsolete NCT alias)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; Waldenstrom macroglobulinemia; prolymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Waldenstrom Macroglobulinemia; Leukemia, Prolymphocytic | interventions — RFB4(dsFv)-PE38 recombinant immunotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BL22 immunotoxin
Procedure: antibody-drug conjugate therapy
Procedure: immunotoxin therapy

SUMMARY:
RATIONALE: BL22 immunotoxin can find tumor cells and kill them without harming normal cells.

PURPOSE: This phase I trial is studying the side effects and best dose of BL22 immunotoxin in treating patients with refractory B-cell chronic lymphocytic leukemia, prolymphocytic leukemia, or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of recombinant BL22 immunotoxin in patients with CD22-positive refractory B-cell chronic lymphocytic leukemia, prolymphocytic leukemia, or indolent non-Hodgkin's lymphoma.
* Determine the safety and efficacy of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the immunogenicity of this drug in these patients.
* Determine the effect of this drug on various components of the circulating cellular immune system in these patients.

OUTLINE: This is a nonrandomized, dose-escalation study. Patients are stratified according to disease type (chronic lymphocytic leukemia vs non-Hodgkin's lymphoma).

Patients receive recombinant BL22 immunotoxin IV over 30 minutes on days 1, 3, and 5. Treatment repeats ≥ every 27 days for up to 6 courses in the absence of neutralizing antibodies to BL22 or PE38, disease progression, or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses beyond CR. Patients who relapse from a CR lasting ≥ 6 months may receive additional courses.

Cohorts of 3-6 patients per stratum receive escalating doses of recombinant BL22 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 24 patients (12 per stratum) will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell leukemia or lymphoma of 1 of the following types:

  * Chronic lymphocytic leukemia

    * Failed standard chemotherapy
  * Prolymphocytic leukemia

    * Failed standard chemotherapy
  * Indolent non-Hodgkin's lymphoma, including mantle cell lymphoma

    * Stage III or IV disease
    * Failed ≥ 1 prior doxorubicin- or fludarabine-containing standard therapy
* CD22-positive disease, as evidenced by 1 of the following:

  * More than 15% malignant cells react with anti-CD22 by immunohistochemistry
  * More than 30% malignant cells are CD22-positive by fluorescence-activated cell sorting analysis
  * More than 400 CD22 sites per malignant cell (average) by radiolabeled anti-CD22 binding
* Treatment is medically indicated, as evidenced by any of the following:

  * Progressive disease-related symptoms
  * Progressive cytopenias due to marrow involvement
  * Progressive or painful splenomegaly or adenopathy
  * Rapidly increasing lymphocytosis
  * Autoimmune hemolytic anemia or thrombocytopenia
  * Increased frequency of infections
* No neutralizing anti-toxin or anti-mouse immunoglobulin G (IgG) antibodies to BL22 or PE38

  * No serum neutralization of > 75% of the activity of 1 μg/mL of BL22
* No CNS disease requiring treatment
* No hairy cell leukemia

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3*
* Platelet count > 40,000/mm^3 NOTE: *Patients with leukemia are eligible regardless of absolute neutrophil count; Grade III-IV pancytopenia or growth factor dependence allowed if due to disease

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* ALT and AST < 2.5 times ULN

Renal

* Creatinine ≤ 1.5 mg/dL

Pulmonary

* FEV1 ≥ 60% of predicted
* DLCO ≥ 55% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior bone marrow transplantation allowed
* More than 3 weeks since prior biologic therapy, including interferon, denileukin diftitox, or LMB-2 immunotoxin
* More than 3 months since prior monoclonal antibody therapy (e.g., rituximab)

Chemotherapy

* See Disease Characteristics
* More than 3 weeks since prior cytotoxic chemotherapy

Endocrine therapy

* More than 1 week since prior steriods

  * Less than 5 doses for non-treatment reasons (e.g., allergy prophylaxis)
  * No evidence of disease response

Radiotherapy

* More than 3 weeks since prior whole-body electron beam radiotherapy

  * Radiotherapy within the past 3 weeks allowed provided the volume of bone marrow treated is < 10% AND the patient has measurable disease located outside the radiation port

Surgery

* Not specified

Other

* More than 3 weeks since prior retinoids
* More than 3 weeks since other prior systemic therapy for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

REFERENCES:
- [Result] Kreitman RJ, Squires DR, Stetler-Stevenson M, Noel P, FitzGerald DJ, Wilson WH, Pastan I. Phase I trial of recombinant immunotoxin RFB4(dsFv)-PE38 (BL22) in patients with B-cell malignancies. J Clin Oncol. 2005 Sep 20;23(27):6719-29. doi: 10.1200/JCO.2005.11.437. Epub 2005 Aug 1. PMID 16061911